CLINICAL TRIAL: NCT01965431
Title: Thorough QT Study to Evaluate the Effects of BI 207127 (Deleobuvir) Combined With Faldaprevir on Cardiac Safety Parameters in Healthy Female and Male Subjects. Randomised, Placebo Controlled, Single-blind, Three-period Crossover Phase-I-study With Moxifloxacin as Positive Control
Brief Title: Thorough QT Study to Evaluate the Effects of BI 207127 (Deleobuvir) Combined With Faldaprevir on Cardiac Safety Parameters in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1241.40; 2013-002741-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — deleobuvir; faldaprevir; Moxifloxacin

ARMS (3):
- BI 207127 + Faldaprevir (Experimental): Tablets/capsules
  Interventions: Drug: BI 207127; Drug: Faldaprevir
- Moxifloxacin (Avalox®) (Active Comparator): Tablets
  Interventions: Drug: Moxifloxacin (Avalox®)
- BI 207127 placebo + Faldaprevir placebo (Experimental): Tablets/capsules
  Interventions: Drug: BI 207127 placebo; Drug: Faldaprevir placebo

INTERVENTIONS:
Drug: BI 207127 — Medium dose oral administration
  Arms: BI 207127 + Faldaprevir
Drug: BI 207127 placebo
  Arms: BI 207127 placebo + Faldaprevir placebo
Drug: Faldaprevir placebo
  Arms: BI 207127 placebo + Faldaprevir placebo
Drug: Faldaprevir — Medium dose oral administration
  Arms: BI 207127 + Faldaprevir
Drug: Moxifloxacin (Avalox®)
  Arms: Moxifloxacin (Avalox®)

SUMMARY:
The objective of this study is to evaluate the effect of multiple doses of BI 207127 combined with faldaprevir on cardiac safety parameters in healthy subjects

ELIGIBILITY:
Inclusion criteria:

* Healthy male and female subjects
* Subjects must be able to understand and comply with study requirements
* Age =18 and =55 years
* BMI range: =18.5 and =29.9 kg/m2

Exclusion criteria:

- any relevant deviation from healthy conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.40.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After an initial screening (Visit 1) within Day -23 and Day -3 prior of the first treatment period, subjects meeting all inclusion and none of the exclusion criteria participated in Visits 2 to 5.
Groups:
- T/R1/R2: Patients were treated with oral dose, started in period 1 with BI 207127 plus Faldaprevir (T) for three days (day -2, -1 and 1): BI 207127 film coated tablets 600 mg (3x200 mg) twice daily (bid) were administered on day -2 and day -1 and 600 mg once daily (qd) on day 1 plus Faldaprevir soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg once daily (qd) on day -1 and day 1 with 240 mL of water, followed in period 2 by matching placebos (R1) for three days (day -2, -1 and 1): matching placebo (BI 207127) three tablets, twice daily (bid) were administered on day -2 and day -1 and three tablets, once daily (qd) on day 1, plus matching placebo (Faldaprevir) soft gelatin two capsules qd on day -2 and one capsule qd on day -1 and day 1 with 240 mL of water, and in period 3 by Moxifloxacin (R2) : Moxifloxacin film coated tablet 400 mg was administered as single dose on day 1 with 240 mL of water. Treatment periods were separated by a wash-out phase of at least 8 days.
- T/R2/R1: Patients were treated with oral dose, started in period 1 with BI 207127 plus Faldaprevir (T) for three days (day -2, -1 and 1): BI 207127 film coated tablets 600 mg (3x200 mg) bid were administered on day -2 and day -1 and 600 mg qd on day 1 plus Faldaprevir soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and day 1 with 240 mL of water, followed in period 2 by Moxifloxacin (R2): Moxifloxacin film coated tablet 400 mg was administered as single dose on day 1 with 240 mL of water, and in period 3 by matching placebos (R1) for three days (day -2, -1 and 1): matching placebo (BI 207127) three tablets, twice daily (bid) were administered on day -2 and day -1 and three tablets, once daily (qd) on day 1, plus matching placebo (Faldaprevir) soft gelatin two capsules qd on day -2 and one capsule qd on day -1 and day 1 with 240 mL of water. Treatment periods were separated by a wash-out phase of at least 8 days.
- R1/T/R2: Patients were treated with oral dose, started in period 1 with matching placebos (R1) for three days (day -2, -1 and 1): matching placebo (BI 207127) three tablets, twice daily (bid) were administered on day -2 and day -1 and three tablets, once daily (qd) on day 1, plus matching placebo (Faldaprevir) soft gelatin two capsules qd on day -2 and one capsule qd on day -1 and day 1 with 240 mL of water, followed in period 2 by BI 207127 plus Faldaprevir (T) for three days (day -2, -1 and 1): BI 207127 film coated tablets 600 mg (3x200 mg) bid were administered on day -2 and day -1 and 600 mg qd on day 1 plus Faldaprevir soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and day 1 with 240 mL of water, and in period 3 by Moxifloxacin (R2):Moxifloxacin film coated tablet 400 mg was administered as single dose on day 1 with 240 mL of water. Treatment periods were separated by a wash-out phase of at least 8 days.
- R1/R2/T: Patients were treated in the morning with oral dose, started in period 1 with matching placebos (R1) for three days (day -2, -1 and 1): matching placebo (BI 207127) three tablets, twice daily (bid) were administered on day -2 and day -1 and three tablets, once daily (qd) on day 1, plus matching placebo (Faldaprevir) soft gelatin two capsules qd on day -2 and one capsule qd on day -1 and day 1 with 240 mL of water, followed in period 2 by Moxifloxacin (R2): Moxifloxacin film coated tablet 400 mg was administered as single dose on day 1 with 240 mL of water, and in period 3 by BI 207127 plus Faldaprevir (T) for three days (day -2, -1 and 1): BI 207127 film coated tablets 600 mg (3x200 mg) bid were administered on day -2 and day -1 and 600 mg qd on day 1 plus Faldaprevir soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and day 1 with 240 mL of water. Treatment periods were separated by a wash-out phase of at least 8 days.
- R2/T/R1: Patients were treated in the morning with oral dose, started in period 1 with Moxifloxacin (R2): Moxifloxacin film coated tablet 400 mg was administered on as single dose on day 1 with 240 mL of water, followed in period 2 by BI 207127 plus Faldaprevir (T) for three days (day -2, -1 and 1): BI 207127 film coated tablets 600 mg (3x200 mg) bid were administered on day -2 and day -1 and 600 mg qd on day 1 plus Faldaprevir soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and day 1 with 240 mL of water, and in period 3 by matching placebos (R1) for three days (day -2, -1 and 1): matching placebo (BI 207127) three tablets, twice daily (bid) were administered on day -2 and day -1 and three tablets, once daily (qd) on day 1, plus matching placebo (Faldaprevir) soft gelatin two capsules qd on day -2 and one capsule qd on day -1 and day 1 with 240 mL of water. Treatment periods were separated by a wash-out phase of at least 8 days.
- R2/R1/T: Patients were treated in the morning with oral dose, started in period 1 with Moxifloxacin (R2): Moxifloxacin film coated tablet 400 mg was administered as single dose on day 1 with 240 mL of water, followed in period 2 by matching placebos (R1) for three days (day -2, -1 and 1): matching placebo (BI 207127) three tablets, twice daily (bid) were administered on day -2 and day -1 and three tablets, once daily (qd) on day 1, plus matching placebo (Faldaprevir) soft gelatin two capsules qd on day -2 and one capsule qd on day -1 and day 1 with 240 mL of water, and in period 3 by BI 207127 plus Faldaprevir (T) for three days (day -2, -1 and 1): BI 207127 film coated tablets 600 mg (3x200 mg) bid were administered on day -2 and day -1 and 600 mg qd on day 1 plus Faldaprevir soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and day 1 with 240 mL of water. Treatment periods were separated by a wash-out phase of at least 8 days.
Period: Overall Study
Arm/Group | T/R1/R2 | T/R2/R1 | R1/T/R2 | R1/R2/T | R2/T/R1 | R2/R1/T
Started | 8 (Started are actually Treated subjects) | 8 | 8 | 8 | 8 | 8
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 6 | 6 | 6 | 6 | 6 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other than stated above | 6 | 5 | 6 | 6 | 6 | 6

BASELINE CHARACTERISTICS:
Population: Treated Set: All subjects who received at least 1 dose of investigational treatment
Groups:
- Overall Study: This study is randomised, single-blind, 3-period crossover having 3 treatments, BI 207127 and Faldaprevir for 3 days (Days -2 to 1), placebo to BI 207127 plus placebo to Faldaprevir for 3 days (Days -2 to 1) and Moxifloxacin 400 mg as single dose (Day 1).
Arm/Group | Overall Study
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Mean Placebo-corrected QTcN Change From Baseline Between 1 to 24 Hours on Day 1 for the Combination Therapy
Description: Maximum mean placebo-corrected QT interval corrected for heart rate according to a parabolic population model (QTcN) change from baseline between 1 to 24 hours on Day 1 for the combination therapy is estimated.
  QTcN denotes the population heart rate corrected QT interval length, based on a parabolic model. 'Baseline' denotes the mean of the pre-dose ECG measurements prior to (first) dose at Visits 2, 3 or 4, determined separately for each treatment period. 'Global baseline' refers to the mean of all available period baseline values.
Time Frame: 20min,15min and 10min prior to drug administration on day -2 (baseline) and 1h (hours), 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h and 24h after drug adminstration on day 1
Population: Electrocardiogram (ECG) analysis set (ECGS): all subjects in the treated set who had at least 1 baseline and post-baseline assessment for at least 1 ECG endpoint.
Measure: Mean (Standard Error); unit: ms
Groups:
- BI 207127+ Faldaprevir: Orally administered BI 207127 film coated tablets 600 mg (3x200 mg) bid on day -2 and day -1 and 600 mg qd on day 1 plus Faldaprevir soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and day 1 with 240 mL of water.
- Placebo to BI 207127 + Placebo to Faldaprevir: Orally administered matching placebo (BI 207127) tablets 600 mg (3x200 mg) bid on day -2 and day -1 and 600 mg qd on day 1 plus matching placebo (Faldaprevir) soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and day 1 with 240 mL of water.
Arm/Group | BI 207127+ Faldaprevir | Placebo to BI 207127 + Placebo to Faldaprevir
Number analyzed (Participants) | 31 | 32
ms | -0.47 (1.65) | -8.37 (1.64)
Statistical Analysis 1: Comparison: BI 207127+ Faldaprevir vs Placebo to BI 207127 + Placebo to Faldaprevir; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is the maximum acceptable extent of statistical and clinical noninferiority of an experimental treatment. Non-inferiority margin for this trial is 10ms; Mean Difference (Net) = 7.90, 90% CI 2-sided [5.37 to 10.43], Standard Error of Mean 1.52 — Maximum mean difference to placebo is estimated. Adjusted means are based on a mixed model for repeated measures with 'global' & 'period-global baseline' covariates. Toeplitz covariance model used for modelling the random and repeated effect

2. Secondary Outcome: Maximum Mean Placebo-corrected QTcN Change From Baseline Between 1 to 6 Hours on Day 1 for the Moxifloxacin Treatment
Description: Maximum mean placebo-corrected QTcN change from baseline between 1 to 6 hours on Day 1 for the Moxifloxacin treatment is estimated.
  QTcN denotes the population heart rate corrected QT interval length, based on a parabolic model. 'Baseline' denotes the mean of the pre-dose ECG measurements prior to (first) dose at Visits 2, 3 or 4, determined separately for each treatment period. 'Global baseline' refers to the mean of all available period baseline values.
Time Frame: 20min,15min and 10min prior to drug administration on day -2 (baseline) and 1h (hours), 2h, 3h, 4h, 5h and 6h after drug adminstration on day 1
Population: ECG analysis set (ECGS)
Measure: Mean (Standard Error); unit: ms
Groups:
- Moxifloxacin: Orally administered Moxifloxacin film coated tablet 400 mg as single dose on day 1 with 240 mL of water.
Arm/Group | Moxifloxacin | Placebo to BI 207127 + Placebo to Faldaprevir
Number analyzed (Participants) | 31 | 32
ms | 14.95 (1.84) | 2.25 (1.74)
Statistical Analysis 1: Comparison: Moxifloxacin vs Placebo to BI 207127 + Placebo to Faldaprevir; No formal hypothesis testing was done; Test type: Superiority or Other; Mean Difference (Net) = 12.70, 90% CI 2-sided [9.32 to 16.08], Standard Error of Mean 2.02 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Maximum Mean Placebo-corrected HR Change From Baseline Between 1 to 24 Hours on Day 1 for the Combination Therapy
Description: Maximum mean placebo-corrected heart rate (HR) change from baseline between 1 to 24 hours on Day 1 for the combination therapy is estimated. HR was derived from the RR interval.
Time Frame: as for outcome 1
Population: ECG analysis set (ECGS)
Measure: Mean (Standard Error); unit: bpm
Groups:
- BI 207127 + Faldaprevir: Orally administered BI 207127 film coated tablets 600 mg (3x200 mg) bid on day -2 and day -1 and 600 mg qd on day 1 plus Faldaprevir soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and day 1 with 240 mL of water.
- Placebo to BI 207127) + Placebo to Faldaprevir: Orally administered matching placebo (BI 207127) tablets 600 mg (3x200 mg) bid on day -2 and day -1 and 600 mg qd on day 1 plus matching placebo (Faldaprevir) soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and day 1 with 240 mL of water.
Arm/Group | BI 207127 + Faldaprevir | Placebo to BI 207127) + Placebo to Faldaprevir
Number analyzed (Participants) | 31 | 32
bpm | -3.47 (0.88) | -3.64 (0.88)
Statistical Analysis 1: Comparison: BI 207127 + Faldaprevir vs Placebo to BI 207127) + Placebo to Faldaprevir; No formal hypothesis testing was done; Test type: Superiority or Other; Mean Difference (Net) = 0.17, 90% CI 2-sided [-1.38 to 1.73], Standard Error of Mean 0.94 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Minimum Mean Placebo-corrected HR (Heart Rate) Change From Baseline Between 1 to 24 Hours on Day 1 for the Combination Therapy
Description: Minimum mean placebo-corrected HR (heart rate) change from baseline between 1 to 24 hours on Day 1 for the combination therapy is estimated. HR was derived from the RR interval.
Time Frame: as for outcome 1
Population: ECG analysis set (ECGS)
Measure: Mean (Standard Error); unit: bpm
Arm/Group | BI 207127 + Faldaprevir | Placebo to BI 207127 + Placebo to Faldaprevir
Number analyzed (Participants) | 31 | 32
bpm | -0.68 (0.88) | 3.74 (0.87)
Statistical Analysis 1: Comparison: BI 207127 + Faldaprevir vs Placebo to BI 207127 + Placebo to Faldaprevir; No formal hypothesis testing was done; Test type: Superiority or Other; Mean Difference (Net) = -4.42, 90% CI 2-sided [-5.98 to -2.87], Standard Error of Mean 0.94 — Minimum mean difference to placebo is estimated. Adjusted means are based on a mixed model for repeated measures with 'global' & 'period-global baseline' covariates. Toeplitz covariance model used for modelling the random and repeated effect

ADVERSE EVENTS:
Time Frame: From the first drug administration until 8 days after the last drug administration, upto 9 days for Moxifloxacin and upto 11 days for BI 207127 + Faldaprevir and Placebo.
Groups:
- BI 207127 + Faldaprevir: Orally administered BI 207127 film coated tablets 600 mg (3x200 mg) bid on day -2 and day -1 and 600 mg qd on day 1 plus Faldaprevir soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and 1 with 240 mL of water.
- Moxifloxacin: Orally administered Moxifloxacin film coated tablet 400 mg as single dose on day1 with 240 mL of water.
- Placebo (BI 207127) + Placebo (Faldaprevir): Orally administered matching placebo (BI 207127) tablets 600 mg (3x200 mg) bid on day -2 and day -1 and 600 mg qd on day 1 plus matching placebo (Faldaprevir) soft gelatin capsules 240 mg (2x120 mg) on day -2 and 120 mg qd on day -1 and 1 with 240 mL of water.
Arm/Group | BI 207127 + Faldaprevir | Moxifloxacin | Placebo (BI 207127) + Placebo (Faldaprevir)
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 17/32 | 4/31 | 7/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 207127 + Faldaprevir (N=32) | Moxifloxacin (N=31) | Placebo (BI 207127) + Placebo (Faldaprevir) (N=32)
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3
Headache (Nervous system disorders) | 10 | 0 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes